CLINICAL TRIAL: NCT05594511
Title: Immediate Effects of the Mandibular Muscle Energy Technique in Patients With Mandibular Joint Pathology and Bruxism. Randomized Controlled Clinical Trial
Brief Title: Mandibular Muscle Energy Technique in Patients With Mandibular Joint Pathology and Bruxism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salamanca (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Principal Investigator, Roberto Méndez Sánchez, Professor, PhD, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-11-386-USalamanca
Record Dates: First submitted 2022-10-20; First posted 2022-10-26 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Temporomandibular Joint Disorders; Bruxism; Pain Threshold; Kinesiophobia
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bruxism; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: randomized, controlled, prospective, double-blind, clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will be blinded because in both groups they were following the treatment and medical recommendations and they will also be attended by a physiotherapist, in one case the mandibular muscular energy technique will be performed and in the other the placebo technique.
  The evaluators did not know to which group the participants belonged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (muscle-energy technique) (Experimental): Mandibular muscle energy technique: In the supine position, the patient will open the mouth and perform isometric contractions for closure controlled by the physiotherapist. Passively, the physiotherapist will increase the range of mandibular opening. The technique consists of performing 3 sets, with 3 isometric contractions in each set of 3 seconds each. At the end of each set, the physiotherapist will passively try to gain mouth opening in order to continue the rest of the sets. At the end of all sets, gently return to the resting position.
  Interventions: Procedure: Muscle-energy mandibular technique
- Control Group (sham technique) (Sham Comparator): Sham technique: In the supine position, the physiotherapist will place his hands under the patient's skull with the fingertips in contact with the suboccipital musculature for 5 minutes, without applying pressure or therapeutic intent. The objective is to provide a stimulus as similar as possible to the original Suboccipital Inhibition Technique, but without force of movement. The patient will keep the eyes closed for the duration of the technique.
  Interventions: Procedure: Sham technique

INTERVENTIONS:
Procedure: Muscle-energy mandibular technique — A single session will be used with the mandibular musculoenergy technique. It will last approximately 2-3 minutes and will be performed by a physiotherapist.
  Arms: Experimental Group (muscle-energy technique)
Procedure: Sham technique — A single session with a sham technique simulating the suboccipital muscle inhibition technique will be used. It will last approximately 2-3 minutes and will be performed by a physiotherapist.
  Arms: Control Group (sham technique)

SUMMARY:
This is a randomized, controlled, double-blind clinical trial. The main objective is to evaluate the immediate effect of the mandibular muscle-energy technique on pain, functionality and kinesiophobia in subjects suffering from temporomandibular dysfunction and bruxism.

In the experimental group the jaw muscle-energy technique will be applied and in the control group a placebo technique will be applied. The intention is to see the immediate effects of the intervention and two evaluations of the pre- and post-intervention outcome variables and a follow-up of kinesiophobia one week later will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study by signing the informed consent form.
* Patients attending maxillofacial consultation with pain, temporomandibular dysfunction and bruxism.
* Pain of at least 3 months of evolution.

Exclusion Criteria:

* Patients with congenital malformations or cervical spine pathology.
* Infectious or inflammatory disease in its acute phase.
* Patients with vertigo or vestibular alterations.
* If there is a contraindication to the technique or phobia on the part of the patient.
* Physiotherapy treatment (manual therapy or electrotherapy) in the last month before their incorporation in the study.
* Pharmacological treatment (analgesics, relaxants and anti-inflammatory drugs) in the last 24 hours before the initial evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-06-23 (Estimated); Study Completion 2023-06-23 (Estimated)

PRIMARY OUTCOMES:
Changes in craniofacial pain intensity | 2 evaluations, one pre-intervention and one post-intervention, 5 minutes after the end of the intervention according to the assigned group.
  For the subjective evaluation of craniofacial pain, the visual analog scale (VAS) will be applied. Scale from 0 (no pain at all) to 10 (maximum possible pain).

SECONDARY OUTCOMES:
Changes in mouth opening mobility | 2 evaluations, one pre-intervention and one post-intervention, 5 minutes after the end of the intervention according to the assigned group.
  The active opening of the mouth will be measured using a digital caliper
Changes in rightward mandibular translation | 2 evaluations, one pre-intervention and one post-intervention, 5 minutes after the end of the intervention according to the assigned group.
  The active rightward mandibular translation will be measured using a digital caliper
Changes in leftward mandibular translation | 2 evaluations, one pre-intervention and one post-intervention, 5 minutes after the end of the intervention according to the assigned group.
  The active leftward mandibular translation will be measured using a digital caliper
Changes in Pressure pain threshold at myofascial trigger point (PT1) of the both upper trapezius muscles | 2 evaluations, one pre-intervention and one post-intervention, 5 minutes after the end of the intervention according to the assigned group.
  The pressure threshold will be recorded using a digital algometer
Changes in pressure pain threshold at myofascial trigger point of the both external pterygoid muscles | 2 evaluations, one pre-intervention and one post-intervention, 5 minutes after the end of the intervention according to the assigned group.
  The pressure threshold will be recorded using a digital algometer
Changes in pressure pain threshold at myofascial trigger point of the both digastric muscles | 2 evaluations, one pre-intervention and one post-intervention, 5 minutes after the end of the intervention according to the assigned group.
  The pressure threshold will be recorded using a digital algometer
Changes in kinesiophobia | 2 evaluations, one pre-intervention and one post-intervention, 5 minutes after the end of the intervention according to the assigned group. And a follow-up after one week
  The Kinesiophobia will be recorded using the spanish version of the Tampa Scale for Kinesiophobia for Temporomandibular Disorders (TSK-TMD-S). It is a valid and reliable instrument for measuring kinesiophobia in patients with TMD, and it uses a Likert scale (1-4) containing 11 items in 2 domains, with higher scores indicating higher levels of kinesiophobia (0-44).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Méndez-Sánchez, PhD, Principal Investigator — University of Salamanca; Antonio Márquez-Vera, PT, Principal Investigator — Institute for Biomedical Research of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No